CLINICAL TRIAL: NCT02961244
Title: Effect of Standard Normothermia Protocol On Surgical Site Infections: Randomized Controlled Trial
Brief Title: Effect of Standard Normothermia Protocol On Surgical Site Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Ali Kadir Değirmenci, Asistant Investigator, MD, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 870-GOA
Record Dates: First submitted 2016-11-01; First posted 2016-11-10 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Surgical Site Infection
Keywords: Surgical Site Infection; normothermia; hypothermia; prewarming
MeSH Terms: conditions — Surgical Wound Infection; Hypothermia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): Perioperative management and warming was not performed according to a standard normothermia protocol, with our clinic's traditional methods except prewarming.
- Intervention Group (Active Comparator): Perioperative management and warming was performed according to a standard normothermia protocol with active prewarming.
  Interventions: Other: Prewarming and perioperative warming with Forced Air Warming device and its blankets.; Device: Forced Air Warming blanket

INTERVENTIONS:
Other: Prewarming and perioperative warming with Forced Air Warming device and its blankets.
  Arms: Intervention Group
Device: Forced Air Warming blanket
  Arms: Intervention Group

SUMMARY:
Aim of this study is to investigate the efficiency of a standard normothermia protocol and effects on postoperative Surgical Site Infection (SSI) rate.

ELIGIBILITY:
Inclusion Criteria:

* Elective
* Preoperatively not infected/dirty Surgical Site
* Open major abdominal operations (hepatobiliary, upper gastrointestinal or colorectal); under general anesthesia, longer than 30 minutes)

Exclusion Criteria:

* Emergent surgery
* Local/locoregional procedures
* Laparoscopic operation
* Minor abdominal operations (e.g. hernia repair, colostomy closure)
* Malign hyperthermia
* Signs of active infection or fever
* Immunosuppression
* Severe malnutrition
* Kidney/liver failure and antibiotic use within the previous 1 week or immunosuppressive use (chemotherapy, steroids.) within the previous 1 month and reversal of patients opinion while randomization period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Cem Terzi, Proffessor Doctor, Study Director — Dokuz Eylul School of Medicine, General Surgery, Colorectal and Pelvic Diseases Department

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Torossian A. Thermal management during anaesthesia and thermoregulation standards for the prevention of inadvertent perioperative hypothermia. Best Pract Res Clin Anaesthesiol. 2008 Dec;22(4):659-68. doi: 10.1016/j.bpa.2008.07.006. PMID 19137809
- [Background] Sessler DI. Perioperative thermoregulation. Geriatr Anesthesiol. 2008;6736(15):107-22
- [Background] Horosz B, Malec-Milewska M. Inadvertent intraoperative hypothermia. Anaesthesiol Intensive Ther. 2013 Jan-Mar;45(1):38-43. doi: 10.5603/AIT.2013.0009. PMID 23572308
- [Background] Doufas AG. Consequences of inadvertent perioperative hypothermia. Best Pract Res Clin Anaesthesiol. 2003 Dec;17(4):535-49. doi: 10.1016/s1521-6896(03)00052-1. PMID 14661656
- [Background] Clinical practice guideline: The management of inadvertent perioperative hypothermia in adults National Collaborating Centre for Nursing and Supportive Care commissioned by National Institute for Health and Clinical Excellence. 2008;88-92, 204-445
- [Background] Putzu M, Casati A, Berti M, Pagliarini G, Fanelli G. Clinical complications, monitoring and management of perioperative mild hypothermia: anesthesiological features. Acta Biomed. 2007 Dec;78(3):163-9. PMID 18330074
- [Background] Reynolds L, Beckmann J, Kurz A. Perioperative complications of hypothermia. Best Pract Res Clin Anaesthesiol. 2008 Dec;22(4):645-57. doi: 10.1016/j.bpa.2008.07.005. PMID 19137808
- [Background] Leslie K, Sessler DI. Perioperative hypothermia in the high-risk surgical patient. Best Pract Res Clin Anaesthesiol. 2003 Dec;17(4):485-98. doi: 10.1016/s1521-6896(03)00049-1. PMID 14661653
- [Background] Torossian A, Brauer A, Hocker J, Bein B, Wulf H, Horn EP. Preventing inadvertent perioperative hypothermia. Dtsch Arztebl Int. 2015 Mar 6;112(10):166-72. doi: 10.3238/arztebl.2015.0166. PMID 25837741
- [Background] Kurz A. Thermal care in the perioperative period. Best Pract Res Clin Anaesthesiol. 2008 Mar;22(1):39-62. doi: 10.1016/j.bpa.2007.10.004. PMID 18494388
- [Background] Leslie K, Sessler DI, Bjorksten AR, Moayeri A. Mild hypothermia alters propofol pharmacokinetics and increases the duration of action of atracurium. Anesth Analg. 1995 May;80(5):1007-14. doi: 10.1097/00000539-199505000-00027. PMID 7726398
- [Background] Fritz HG, Holzmayr M, Walter B, Moeritz KU, Lupp A, Bauer R. The effect of mild hypothermia on plasma fentanyl concentration and biotransformation in juvenile pigs. Anesth Analg. 2005 Apr;100(4):996-1002. doi: 10.1213/01.ANE.0000146517.17910.54. PMID 15781513
- [Background] Polderman KH. Mechanisms of action, physiological effects, and complications of hypothermia. Crit Care Med. 2009 Jul;37(7 Suppl):S186-202. doi: 10.1097/CCM.0b013e3181aa5241. PMID 19535947
- [Background] Liu M, Hu X, Liu J. The effect of hypothermia on isoflurane MAC in children. Anesthesiology. 2001 Mar;94(3):429-32. doi: 10.1097/00000542-200103000-00011. PMID 11374601
- [Background] Mauermann WJ, Nemergut EC. The anesthesiologist's role in the prevention of surgical site infections. Anesthesiology. 2006 Aug;105(2):413-21; quiz 439-40. doi: 10.1097/00000542-200608000-00025. No abstract available. PMID 16871076
- [Background] Kurz A, Sessler DI, Lenhardt R. Perioperative normothermia to reduce the incidence of surgical-wound infection and shorten hospitalization. Study of Wound Infection and Temperature Group. N Engl J Med. 1996 May 9;334(19):1209-15. doi: 10.1056/NEJM199605093341901. PMID 8606715
- [Background] Wenisch C, Narzt E, Sessler DI, Parschalk B, Lenhardt R, Kurz A, Graninger W. Mild intraoperative hypothermia reduces production of reactive oxygen intermediates by polymorphonuclear leukocytes. Anesth Analg. 1996 Apr;82(4):810-6. doi: 10.1097/00000539-199604000-00023. PMID 8615502
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for prevention of surgical site infection, 1999. Hospital Infection Control Practices Advisory Committee. Infect Control Hosp Epidemiol. 1999 Apr;20(4):250-78; quiz 279-80. doi: 10.1086/501620. No abstract available. PMID 10219875
- [Background] Barie PS. Surgical site infections: epidemiology and prevention. Surg Infect (Larchmt). 2002;3 Suppl 1:S9-21. doi: 10.1089/sur.2002.3.s1-9. PMID 12573036
- [Background] Arslan NC, Terzi C, Kaya Ozlem, et. al. Perioperative Body Temperature: One Day Prevalence Study İn One Hospital. XVI. Annual Meeting of the European Society of Surgery Abstract Book 2012; 667-886
- [Background] Byrne DJ, Malek MM, Davey PG, Cuschieri A. Postoperative wound scoring. Biomed Pharmacother. 1989;43(9):669-73. doi: 10.1016/0753-3322(89)90085-1. PMID 2696565
- [Background] Horan TC, Gaynes RP, Martone WJ, Jarvis WR, Emori TG. CDC definitions of nosocomial surgical site infections, 1992: a modification of CDC definitions of surgical wound infections. Infect Control Hosp Epidemiol. 1992 Oct;13(10):606-8. No abstract available. PMID 1334988
- [Background] Bratzler DW, Dellinger EP, Olsen KM, Perl TM, Auwaerter PG, Bolon MK, Fish DN, Napolitano LM, Sawyer RG, Slain D, Steinberg JP, Weinstein RA; American Society of Health-System Pharmacists; Infectious Disease Society of America; Surgical Infection Society; Society for Healthcare Epidemiology of America. Clinical practice guidelines for antimicrobial prophylaxis in surgery. Am J Health Syst Pharm. 2013 Feb 1;70(3):195-283. doi: 10.2146/ajhp120568. No abstract available. PMID 23327981
- [Background] Culver DH, Horan TC, Gaynes RP, Martone WJ, Jarvis WR, Emori TG, Banerjee SN, Edwards JR, Tolson JS, Henderson TS, et al. Surgical wound infection rates by wound class, operative procedure, and patient risk index. National Nosocomial Infections Surveillance System. Am J Med. 1991 Sep 16;91(3B):152S-157S. doi: 10.1016/0002-9343(91)90361-z. PMID 1656747
- [Background] Elixhauser A, Steiner C, Harris DR, Coffey RM. Comorbidity measures for use with administrative data. Med Care. 1998 Jan;36(1):8-27. doi: 10.1097/00005650-199801000-00004. PMID 9431328
- [Background] Forbes SS, Eskicioglu C, Nathens AB, Fenech DS, Laflamme C, McLean RF, McLeod RS; Best Practice in General Surgery Committee, University of Toronto. Evidence-based guidelines for prevention of perioperative hypothermia. J Am Coll Surg. 2009 Oct;209(4):492-503.e1. doi: 10.1016/j.jamcollsurg.2009.07.002. Epub 2009 Aug 20. No abstract available. PMID 19801323
- [Background] Thiele RH, Huffmyer JL, Nemergut EC. The "six sigma approach" to the operating room environment and infection. Best Pract Res Clin Anaesthesiol. 2008 Sep;22(3):537-52. doi: 10.1016/j.bpa.2008.06.002. PMID 18831302
- [Background] Sessler DI, Schroeder M, Merrifield B, Matsukawa T, Cheng C. Optimal duration and temperature of prewarming. Anesthesiology. 1995 Mar;82(3):674-81. doi: 10.1097/00000542-199503000-00009. PMID 7879936
- [Background] Horn EP, Bein B, Bohm R, Steinfath M, Sahili N, Hocker J. The effect of short time periods of pre-operative warming in the prevention of peri-operative hypothermia. Anaesthesia. 2012 Jun;67(6):612-7. doi: 10.1111/j.1365-2044.2012.07073.x. Epub 2012 Feb 29. PMID 22376088
- [Background] Melling AC, Ali B, Scott EM, Leaper DJ. Effects of preoperative warming on the incidence of wound infection after clean surgery: a randomised controlled trial. Lancet. 2001 Sep 15;358(9285):876-80. doi: 10.1016/S0140-6736(01)06071-8. PMID 11567703
- [Background] Wong PF, Kumar S, Bohra A, Whetter D, Leaper DJ. Randomized clinical trial of perioperative systemic warming in major elective abdominal surgery. Br J Surg. 2007 Apr;94(4):421-6. doi: 10.1002/bjs.5631. PMID 17380549
- [Background] de Brito Poveda V, Clark AM, Galvao CM. A systematic review on the effectiveness of prewarming to prevent perioperative hypothermia. J Clin Nurs. 2013 Apr;22(7-8):906-18. doi: 10.1111/j.1365-2702.2012.04287.x. Epub 2012 Sep 17. PMID 22978458
- [Background] Llewellyn L. Effect of Pre-warming on Reducing the Incidence of Inadvertent Peri-operative Hypothermia for Patients Undergoing General Anaesthesia: A Mini-review. Br J Anaesth Recover Nurs. 2013;14(1-2):3-10
- [Background] Flores-Maldonado A, Medina-Escobedo CE, Rios-Rodriguez HM, Fernandez-Dominguez R. Mild perioperative hypothermia and the risk of wound infection. Arch Med Res. 2001 May-Jun;32(3):227-31. doi: 10.1016/s0188-4409(01)00272-7. PMID 11395189
- [Background] Barone JE, Tucker JB, Cecere J, Yoon MY, Reinhard E, Blabey RG Jr, Lowenfels AB. Hypothermia does not result in more complications after colon surgery. Am Surg. 1999 Apr;65(4):356-9. PMID 10190363
- [Background] Lehtinen SJ, Onicescu G, Kuhn KM, Cole DJ, Esnaola NF. Normothermia to prevent surgical site infections after gastrointestinal surgery: holy grail or false idol? Ann Surg. 2010 Oct;252(4):696-704. doi: 10.1097/SLA.0b013e3181f6c2a9. PMID 20881777
- [Background] Pu Y, Cen G, Sun J, Gong J, Zhang Y, Zhang M, Wu X, Zhang J, Qiu Z, Fang F. Warming with an underbody warming system reduces intraoperative hypothermia in patients undergoing laparoscopic gastrointestinal surgery: a randomized controlled study. Int J Nurs Stud. 2014 Feb;51(2):181-9. doi: 10.1016/j.ijnurstu.2013.05.013. Epub 2013 Jun 17. PMID 23787221
- [Background] Esnaola NF, Cole DJ. Perioperative normothermia during major surgery: is it important? Adv Surg. 2011;45:249-63. doi: 10.1016/j.yasu.2011.03.007. PMID 21954692
- [Background] Melton GB, Vogel JD, Swenson BR, Remzi FH, Rothenberger DA, Wick EC. Continuous intraoperative temperature measurement and surgical site infection risk: analysis of anesthesia information system data in 1008 colorectal procedures. Ann Surg. 2013 Oct;258(4):606-12; discussion 612-3. doi: 10.1097/SLA.0b013e3182a4ec0f. PMID 23989047

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 2013 and December 2015 elective, preoperatively not infected/dirty, open major abdominal operations under general anesthesia, longer than 30 minutes and over 18 aged were included in the study. Primary outcome was comparison of SSI rates between groups and secondary was effects of protocol to normothermia.
Pre-assignment Details: Exclusion criteria were emergent surgery, local/locoregional procedures, laparoscopic operations, minor abdominal operations, malign hyperthermia, signs of active infection/fever, immunosuppression, malnutrition, kidney/liver failure, antibiotic use within the previous 1 week/ımmunsupresive use within previous 1 month, reversal of approval.
Groups:
- Intervention Group: Perioperative management and warming was performed according to a standard normothermia protocol with active prewarming.
  Prewarming and perioperative warming with Forced Air Warming device and its blankets.
  Forced Air Warming blanket
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 64 | 64
Patients Excluded During Randomization | 0 | 1
Completed | 63 | 55
Not Completed | 1 | 9
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Surgery plan change after study approval | 0 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — İnadequate data | 0 | 2

BASELINE CHARACTERISTICS:
Units Other Than Participants: Patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 63 | 55 | 118
Number analyzed (Patients) | 63 | 55 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] — For age variable, groups were homogeneous. (p=0.870)
  years | 58.0 (14.3) | 57.6 (12.9) | 57.8 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants] — For gender variable, groups were homogeneous. (p=0.190)
  Participants
    Female | 34 | 23 | 57
    Male | 29 | 32 | 61
BMI [Mean (Standard Deviation); unit: kilograms per square meter] — For BMI variable, groups were homogeneous. (p=0.836)
  kilograms per square meter | 26.6 (4.9) | 26.8 (4.4) | 26.7 (4.7)
Weight [Mean (Standard Deviation); unit: kilograms] — For weight variable, groups were homogeneous. (p=0.346)
  kilograms | 72.8 (14.9) | 75.3 (14.5) | 74 (14.7)
Height [Mean (Standard Deviation); unit: centimeters] — For height variable, groups were homogeneous. (p=0.166)
  centimeters | 165.1 (8.6) | 167.3 (8.7) | 166.0 (8.0)
Ethiology [Count of Participants; unit: Participants] — Etiologies including hepatopancreaticobiliary, colorectal, upper gastrointestinal systems diseases .
  Participants
    Hepatopancreaticobiliary System Etiology | 24 | 10 | 34
    Colorectal Tract Etiology | 32 | 32 | 64
    Upper Gastointestinal Tract | 7 | 13 | 20
Smoking habit [Count of Participants; unit: Participants] — For smoking habit both groups were homogenous.(p=0.893)
  Participants
    Nonsmoker | 30 | 26 | 56
    Smoking History | 33 | 29 | 62
Alcohol Use [Count of Participants; unit: Participants] — For alcohol use, groups were homogeneous. (p=0.541)
  Participants
    Alcohol use (<2 glass) | 61 | 52 | 113
    Alcohol use (≥2 glass) | 2 | 3 | 5
Type of anesthesia [Count of Participants; unit: Participants] — For anesthesia choice, groups were homogeneous. (p=0.655)
  Participants
    General anesthesia | 16 | 15 | 31
    General and epidural anesthesia | 29 | 20 | 49
    General and intrathecal anesthesia | 18 | 20 | 38
Epidural catheter removal time if any inserted [Mean (Standard Deviation); unit: days] — For epidural catheher removal time, groups were homogeneous. (p=0.973) Population: For patients only had had epidural catheter inserted.
  days
    number analyzed (Participants) | 29 | 20 | 49
    (all) | 5.07 (2.3) | 5.09 (2) | 5.08 (2.2)
Central venous access [Count of Participants; unit: Participants] — For cetral venous access choice groups were homogeneous. (p=0.107)
  Participants
    Not used | 18 | 21 | 39
    Used temporary methods | 33 | 20 | 53
    Permenant central venous port previously inserted | 12 | 14 | 26
If only temporary, removal time of central venous catheter [Mean (Standard Deviation); unit: days] — For temporary central venous catheter removing time both groups were homogenous. (p=0.259) Population: For patients only had had temporary central venous catheter inserted.
  days
    number analyzed (Participants) | 33 | 20 | 53
    (all) | 6.09 (3.7) | 7.2 (2.6) | 6.5 (3.4)
Operating Room Temperature [Mean (Standard Deviation); unit: ºC degrees] — For operating room temperature variable, groups were homogeneous. (p=0.059)
  ºC degrees | 21.3 (2) | 21.5 (2) | 21.4 (2)
İntraoperative blood loss [Mean (Standard Deviation); unit: liters] — For intraoperative blood loss data, groups were homogeneous. (p=0.614)
  liters | 0.23 (0.3) | 0.26 (0.36) | 0.24 (0.33)
İntraoperative red cell transfusion [Mean (Standard Deviation); unit: units] — For intraoperative red cell transfusion variable, groups were homogeneous. (p=0.470)
  units | 0.24 (0.58) | 0.33 (0.74) | 0.25 (0.6)
Intraoperative fresh frozen plasma transfusion [Mean (Standard Deviation); unit: units] | 0 (0) | 0.018 (0.134) | 0.008 (0.009)
Intraoperative cristalloid fluid [Mean (Standard Deviation); unit: liters] — For cristalloid fluid infusement amounts, groups were homogeneous. (p=0.855)
  liters | 3.06 (1.38) | 3.01 (1.4) | 3.04 (1.38)
Intraoperative colloid fluid [Mean (Standard Deviation); unit: liters] — For colloid fluid infusement amounts, groups were homogeneous. (p=0.361)
  liters | 0.42 (0.57) | 0.33 (0.42) | 0.38 (0.5)
Intraoperative urine output [Mean (Standard Deviation); unit: liters] — For peroperative urine output, groups were homogeneous. (p=0.559)
  liters | 0.77 (0.71) | 0.7 (0.57) | 0.74 (0.64)
Mean heart rate [Mean (Standard Deviation); unit: beats per minute] — For mean heart rate amounts, groups were homogeneous. (p=0.390)
  beats per minute | 78 (13.4) | 75.8 (14.5) | 77 (13.9)
Intraoperative mean arterial blood pressure [Mean (Standard Deviation); unit: mm Hg] — For intraoperative mean arterial blood pressure levels, groups were homogeneous. (p=0.388)
  mm Hg | 89.1 (13.2) | 87 (7) | 88.1 (13.4)
Operation duration [Mean (Standard Deviation); unit: minutes] — For operation duration , groups were homogeneous. (p=0.059)
  minutes | 239.6 (118.3) | 199.9 (106.3) | 221.1 (114)
Perioperative hemoglobin levels [Mean (Standard Deviation); unit: g/dl] — Preoperative (p=0.984), postoperative first day (p=0.526) and ∆(Hemoglobin)(the difference between preoperative and postoperative first day levels)(p=0.385)
  g/dl
    Preoperative | 11.81 (1.49) | 11.8 (1.35) | 11.81 (1.42)
    Postoperative 1. Day | 11.0 (1.58) | 11.19 (1.54) | 11.09 (1.55)
    ∆(Hemoglobin) | 0.80 (1.22) | 0.61 (1.10) | 0.71 (1.16)
Perioperative albumin levels [Mean (Standard Deviation); unit: g/dl] — Preoperative (p=0.359), postoperative first day (p=0.314) and ∆(Albumin)(the difference between preoperative and postoperative first day levels)(p=0.055)
  g/dl
    Preoperative | 3.74 (0.46) | 3.66 (0.5) | 3.71 (0.48)
    Postoperative 1. Day | 2.86 (0.56) | 2.96 (0.5) | 2.91 (0.53)
    ∆(Albumin) | 0.88 (0.51) | 0.69 (0.5) | 0.79 (0.51)
Profilactic antibiotics [Count of Participants; unit: Participants] — There were not enough numbers in all boxes so statistical analyses not appropriate to assess for this title.
  Participants
    Cefazolin | 30 | 22 | 52
    Cefuroxime + metronidazole | 30 | 32 | 62
    Ceftriaxone | 1 | 1 | 2
    Ceftriaxone+ metronidazole | 1 | 0 | 1
    Amoxicillin + clavulanate | 1 | 0 | 1
Duration of Hospitalization Parameters [Mean (Standard Deviation); unit: days] — Between two groups duration of hospitalizations were not statistically different including parameters of Total Duration of Hospitalization (p=0.879), Preoperative Duration of Hospitalization (p=0.601), Postoperative Duration of Hospitalization (0.995) and Duration of ICU Hospitalization (0.346). Population: In our study 11 patients from intervention group and 16 patients from control group needed ICU follow up after surgery. (p=0.348)
  days
    Total Duration of Hospitalization | 18.96 (18.62) | 19.4 (10.49) | 19.25 (15.28)
    Preoperative Duration of Hospitalization | 6.87 (5.91) | 7.47 (6.49) | 7.15 (6.17)
    Postoperative Duration of Hospitalization | 12.09 (15.54) | 12.1 (9.07) | 12.1 (12.88)
    Duration of ICU Hospitalization: number analyzed (Participants) | 16 | 11 | 27
    Duration of ICU Hospitalization | 3.5 (5.68) | 3.45 (7.48) | 3.48 (6.33)
Simple Hospitalization costs [Mean (Standard Deviation); unit: Thousand Turkish liras] — These data is not result of standardized (like in the literature suggests) costs data.These data made by our patients data system which can calculate goverments payments fees, etc for any procedure performed to any patient. (intervention based data ) (p=0.524)
  Thousand Turkish liras | 12.6 (9.8) | 11.7 (6.1) | 12.2 (8.3)
Perioperative Warming [Number; unit: participants] — There were not enough numbers in all boxes so statistical analyses not appropriate to assess for preoperative and peroperative warming. Postoperative warming choices were significiantly different between two groups as excepted because of study protocols contents.(p<0.001) Population: Preoperative Warming which is not our center's traditional method for routine maintaining normothermia procedures, performed for only and to all of intervention group patients . For this reason it is not inculed to this analyze table.
  participants
    Peroperatuar Warming | 63 | 55 | 118
    Postoperative Warming: number analyzed (Participants) | 13 | 55 | 68
    Postoperative Warming | 13 | 47 | 60
Surgical Site Classification [Count of Participants; unit: Participants] — During the preoperative patient's approval period, if surgical site is predicted as contaminated and dirty, these patients not appropriate for study. (preoperatively) In 2 patients preoperatively appropriate was found that peroperatively they had closed microperforation of tumor.Though minimal contamination detected perioperatively and there were not any clinical findings of infection, they accepted as contaminated.
  There were not enough numbers in all boxes so statistical analyses not appropriate to assess.
  Participants
    Clean | 4 | 2 | 6
    Clean-Contaminated | 58 | 52 | 110
    Contaminated | 1 | 1 | 2
ASA Score [Count of Participants; unit: Participants] — For ASA scores groups were homogeneous. (p=0.943) ASA 4,5,6 is not shown because of the study inclusion criterias. (ASA which has known as American Society of Anesthesiologists Physical Status, min. 1 and max. 6). Definitions: ASA 1-Normal healthy patients, ASA 2-A patient with mild systemic disease. ASA 3-A Patient with severe systemic disease, ASA4-A patient with severe systemic disease that is a constant threat to life, ASA5-A moribund patient who is not expected to survive without the operation, ASA6-A declared brain-dead patient whose organs are being removed for donor purposes)
  Participants
    ASA 1 | 22 | 19 | 41
    ASA 2 | 32 | 29 | 61
    ASA 3 | 9 | 7 | 16
NNISS Score [Count of Participants; unit: Participants] — For NNISS scores groups were homogeneous. (p=0.875) NNISS Score which has known as The National Nosocomial Infections Surveillance System Scoring System used for prediction of the risk of Surgical Site İnfections (SSI).The NNIS basic SSI risk index is composed of the following criteria: American Society of Anesthesiologists score of 3, 4, or 5 (>2 takes one score; wound class( contaminated or dirty takes one point; and duration of surgery (There are percantile times defined and above 75 percantile, score takes one point) NNISS Score may be 0 to 3, and SSI risks were increased by score.
  Participants
    <2 | 52 | 46 | 98
    ≥2 | 11 | 9 | 20
SENIC Score [Count of Participants; unit: Participants] — For SENIC scores groups were homogeneous. (0.581) This Scoring system has known as Study on Efficacy of Nosocomial Infection Control (SENIC) project's SSI Risk Scoring System (Min. 0 to max. 4 points may be calculated , risk of SSI incerases by score ). 4 criterias include duration of surgery (>2 hours), abdominal surgery, wound class( contaminated or dirty takes one point) and comorbidities (>2) which is any of them is one points.
  Because of the participants who in each score (0-4) was not enough to analyse statisticaly, participants divided into two groups. (<3 and ≥3)
  Participants
    <3 | 57 | 48 | 105
    ≥3 | 6 | 7 | 13
Comorbidities [Count of Participants; unit: Participants] — There were not enough numbers in all boxes so statistical analyses not appropriate to assess for this title. Buy for classifaciton of the comobidities, Elixhauser Classification used for standart data presentation.
  Participants
    Congestive Heart Failure | 1 | 2 | 3
    Pulmonary Circulation Disorders | 0 | 5 | 5
    Complicated Hypertension | 2 | 4 | 6
    Uncomplicated Hypertension | 19 | 19 | 38
    Chronic Respiratory Diseases | 2 | 4 | 6
    Uncomplicated Diabetes | 11 | 10 | 21
    Complicated Diabetes | 0 | 3 | 3
    Hypothyroidism | 8 | 3 | 11
    Lymphoma | 1 | 1 | 2
    Metastatic Cancer | 16 | 11 | 27
    Non-metastatic Solid Tumor | 45 | 43 | 88
    Other(Valvuler, collagen tissue, etc diseases) | 4 | 1 | 5
Perioperative Temperature Measurements [Mean (Standard Deviation); unit: ºC degrees] — Perioperative Minimum Measurement p<0.001 Preoperative Room Enterance Temperature p=0.980 Preoperative Room Exit Temperature p=0.094 After Entubation Temperature p=0.011 Postentubation 60. minutes Temperature p<0.001 Postentubation 120. minutes Temperature p<0.001 Postentubation 180. minutes Temperature p=0.001 Postentubation 240. minutes Temperature p=0.001 After Extubation Temperature p<0.001 Recovery Room Enterance Temperature p<0.001 Recovery Room ExitTemperature p=0.094 Service Enterance Temperature p=0.716 Population: In our study 11 patients from intervention group and 16 patients from control group needed ICU follow-up after surgery. For this reason ICU patient's measurements were not including service data.
  Also these measurements were not including 300, 360, 420, 480, 540, 600 minutes data.Because most of the patients operation times are less than 6 hours.
  ºC degrees
    Perioperative Minimum Measurement | 35.17 (0.59) | 35.76 (0.52) | 35.44 (0.63)
    Preoperative Room Enterance Temperature | 36.94 (0.47) | 36.94 (0.46) | 36.94 (0.46)
    Preoperative Room Exit Temperature | 37.03 (0.4) | 36.89 (0.5) | 36.96 (0.46)
    After Entubation Temperature | 36.36 (0.6) | 36.66 (0.46) | 36.5 (0.56)
    Postentubation 60. minutes Temperature | 35.74 (0.62) | 36.16 (0.56) | 35.9 (0.62)
    Postentubation 120. minutes Temperature | 35.8 (0.73) | 36.28 (0.6) | 35.9 (0.76)
    Postentubation 180. minutes Temperature | 35.63 (0.86) | 36.25 (0.72) | 35.88 (0.86)
    Postentubation 240. minutes Temperature | 35.5 (0.82) | 36.45 (0.87) | 35.85 (0.95)
    After Extubation Temperature | 35.88 (0.74) | 36.54 (0.67) | 36.21 (0.77)
    Recovery Room Enterance Temperature | 35.84 (0.75) | 36.41 (0.64) | 36.12 (0.75)
    Recovery Room ExitTemperature | 36.48 (0.62) | 36.7 (0.61) | 36.59 (0.62)
    Service Enterance Temperature: number analyzed (Participants) | 47 | 44 | 91
    Service Enterance Temperature | 36.31 (0.42) | 36.35 (0.38) | 36.33 (0.4)
    ICU Enterance Temperature (ICU patients): number analyzed (Participants) | 16 | 11 | 27
    ICU Enterance Temperature (ICU patients) | 35.78 (0.95) | 36.08 (0.64) | 35.89 (0.85)
Infectious Complications [Count of Participants; unit: Participants] — Our study's main outcome which is SSI is significiantly different between two groups.(p=0.044)
  Participants
    No İnfectious Complications | 42 | 43 | 85
    Pulmonary | 4 | 1 | 5
    Urinary | 2 | 2 | 4
    Bacteriemia | 3 | 1 | 4
    SSI | 18 | 9 | 27
SSI Classification [Count of Participants; unit: Participants]
  Superficial Incisional | 10 | 6 | 16
  Deep Incisional | 3 | 1 | 4
  Organ-Space | 5 | 2 | 7
ASEPSIS Total Scores [Mean (Standard Deviation); unit: points] — ASEPSIS Wound Scoring System used in our study. ASEPSIS postoperative total Points (p=0.029) was different between two groups. Simply points are given for the need for Additional treatment, the presence of Serous discharge, Erythema, Purulent exudate, and Separation of the deep tissues, the Isolation of bacteria, and the duration of inpatient Stay (ASEPSIS). (min. is 0 points and max. doesn't have any limit but 0-10 points is succesful, 11-20 points is impaired healing and 21-30 points is mild, 31-40 is moderate, >41 points is severe SSI.)
  points | 17.83 (13.83) | 12.64 (10.6) | 15.41 (12.67)

OUTCOME MEASURES:

1. Primary Outcome: Surgical Site Infection Rate
Description: Within the postoperative 30 days, if there is purulent exudate or nonpurulent but culture was pozitive, we accepted them as Surgical Site Infection (SSI) diagnosed.
  All patients were made enough incision wide to explore their entire abdomen defined as "Major Abdominal Surgery" .
  With this results between two groups intervention group had lesser rates of SSI respectively( (p=0.045 Mann Whitney U, n<30), (p=0.044 chi-square )
Time Frame: Postoperative 30 days
Population: Patients and their results assessed on the basis of intention to treat per protocole.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 63 | 55
Participants | 19 | 8

2. Secondary Outcome: Maintaining Normothermia Rate
Description: Within the surgery day, from patient bed through the operating room to PACU or ICU or back to patient bed.
  With these results our intervention group's maintaining normothermia rates were higher respectively. ( p=0.001) For each patients around 11 temperature measurement had been made according to the operation time . If any measurement of any patients was <36 ºC , that patient accepted as hypothermic. (Failure to maintain normothermia)
Time Frame: Surgery day
Population: Patients and their results assessed on the basis of intention to treat per protocole.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 63 | 55
Participants | 7 | 26

ADVERSE EVENTS:
Time Frame: Within the postoperative 30 days
Arm/Group | Control Group | Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/55
Other Adverse Events (participants affected / at risk) | 0/63 | 1/55
OTHER ADVERSE EVENTS (reported when occurring in more than 0.008% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=63) | Intervention Group (N=55)
Thermal Discomfort (Product Issues) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Surgical etiologies were various.It was a single-centered trial whose power was 80%.The room temperatures could not be kept constant.The number of samples were not enough to make variate analysis of SSI and hypothermia risk factors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No